CLINICAL TRIAL: NCT04219189
Title: The Acute Effect of Vaping on Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Pennington Biomedical Research Center (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HM20018382; 2019-066-PBRC (Other: Pennington Biomedical Research Center); U54DA036105 (NIH)
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Energy Intake; Food Intake; E-Cig Use; Appetite
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: This study consists of a baseline assessment which is followed by two within-subject, laboratory conditions that differ by the product used: 1) JUUL e-cigarette with a 5% nicotine pod, 2) no active e-cigarette use (uncharged JUUL with empty pod). The condition orders (i.e., 1 then 2, or 2 then 1) will be randomly ordered and assigned following enrollment. During the vaping condition, participants will be asked to take 20 e-cigarette puffs over 20 minutes before consuming an ad libitum buffet meal. During the alternative control condition, participants will have access to an uncharged JUUL with an empty pod for 20 minutes (instead of vaping) before consuming an ad libitum buffet meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaping to Control Group (Experimental): Participants in this arm will undergo the vaping condition during the first visit and the control condition during the second visit.
  Interventions: Other: Vaping condition; Other: Control condition
- Control to Vaping Group (Experimental): Participants in this arm will undergo the control condition during the first visit and the vaping condition during the second visit.
  Interventions: Other: Vaping condition; Other: Control condition

INTERVENTIONS:
Other: Vaping condition — Participants will be asked to use a JUUL device to vape 20 puffs over 20 minutes. Participants will use JUUL pods with ~5% nicotine by weight. The anticipated amount of nicotine that will be absorbed with 20 puffs is approximately 1.6 mg, which is equal to approximately 1.5 cigarettes.
Other: Control condition — Participants will have access to an uncharged JUUL device with an empty pod for 20 minutes.

SUMMARY:
This study assesses the acute effects of a standardized 20-minute vaping episode compared to a non-vaping control condition on ad libitum food intake during a 30-minute buffet meal, occurring approximately 45 minutes after the vaping episode

DETAILED DESCRIPTION:
Weight control is a common motive for cigarette smoking and nicotine has been shown to suppress appetite and increase resting metabolic rate, and also serves as a behavioral alternative to eating or a distraction from hunger or food craving. Data on the acute effect of e-cigarette use ('vaping') on ad libitum food intake are non-existent. Given that many e-cigarette users report vaping for weight control and that certain e-cigarettes are being actively marketed for weight management and/or suppression of food cravings, addressing this research gap is of the utmost importance.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age (ID card verified)
* Reports either everyday e-cigarette use with liquid containing at least 0.3% (~3 mg/ml) nicotine or some day e-cigarette use ( at least 3 days a week) with liquid containing at least 3% (~30 mg/ml) nicotine for the past 30 days.

Exclusion Criteria:

* being unwilling to consume the foods provided due to: a) dietary limitations or preferences or b) allergies to the foods provided.
* being unwilling to take 20 puffs from a JUUL device containing a 5% nicotine pod
* self-reported current, diagnosed medical condition(s) will be excluded automatically: heart-related conditions (e.g., recent heart attack/stroke, coronary heart disease), severe immune system disorders (e.g., HIV/AIDS, multiple sclerosis), respiratory disorders (e.g., COPD, asthma), kidney diseases, liver diseases (e.g., cirrhosis), or seizures
* observed high blood pressure at screening (systolic >140; diastolic >90)
* other self-reported current, diagnosed medical conditions (e.g., specific food allergies, diabetes, thyroid disease, lyme disease) will be considered for exclusion after consultation with the PI and medical monitor
* self-reported current, diagnosed psychiatric conditions or who report current psychiatric treatment or psychotropic medication use
* past month use of cocaine, opioids, benzodiazepines, methamphetamine, or other (non-cannabis) illicit drugs
* self-report of >25 days out of the past 30 for alcohol use or >20 days out of the past 30 for cannabis use.
* women who are breast-feeding or test positive for pregnancy (by urinalysis at screening)
* women using progestin-IUDS for birth control
* women using birth control injections (e.g., Depo-Provera)
* women who received a hysterectomy and still have ovaries present
* self-report intending to quit tobacco/nicotine products in the next 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Cobb (Amey), PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Center for the Study of Tobacco Products, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaping to Control Group | Control to Vaping Group
Started | 19 | 21
Completed | 18 | 16
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Participant blood pressure out of range for the study , withdrawn by PI | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaping to Control Group | Control to Vaping Group | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (6.7) | 26.9 (10.1) | 25.7 (8.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 12 | 9 | 21
  Non-Binary | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Middle Eastern | 3 | 1 | 4
  Asian | 1 | 4 | 5
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  Prefer to self describe | 1 | 1 | 2
  White | 8 | 7 | 15
  More than one race | 1 | 2 | 3
  Unknown or not reported | 0 | 0 | 0
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown ethnicity or not reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Energy Intake
Description: Energy intake in kilocalories (kcal) during the ad libitum buffet meal will be measured via directly weighed food provision and waste (food/energy intake is calculated by difference).
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: Kilocalories
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
Kilocalories
  Kilocalories (active ) | 1102.1 (615.3) | 1003.4 (577.5)
  Kilocalories (control) | 910.4 (529.4) | 868.3 (443.6)

2. Secondary Outcome: Dietary Added Sugar Intake
Description: Dietary added sugar intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
grams
  Added Sugar (active) | 28.4 (27.5) | 43.0 (28.9)
  Added sugar (control) | 25.0 (19.7) | 37.7 (24.4)

3. Secondary Outcome: Dietary Sugar Intake
Description: Dietary sugar intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
grams
  Sugar (active) | 32.9 (28.0) | 54.0 (41.3)
  Sugar (control) | 29.2 (20.1) | 50.0 (38.0)

4. Secondary Outcome: Dietary Fat Intake
Description: Dietary fat intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
grams
  Fat (active) | 40.9 (27.6) | 52.9 (27.6)
  Fat (control) | 37.7 (24.3) | 51.2 (28.4)

5. Secondary Outcome: Dietary Carbohydrate Intake
Description: Dietary carbohydrate intake
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
grams
  Carb (active) | 82.2 (51.8) | 106.6 (62.0)
  Carb (control) | 72.8 (34.8) | 105.3 (55.1)

6. Secondary Outcome: Dietary Protein Intake
Description: Dietary protein intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
grams
  Protein (active) | 51.7 (33.7) | 58.3 (34.1)
  Protein (control) | 46.7 (29.0) | 53.1 (34.1)

7. Secondary Outcome: Dietary Calcium Intake
Description: Dietary calcium intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
milligrams
  Calcium (active) | 287.1 (332.5) | 404.5 (269.8)
  Calcium (control) | 294.4 (294.9) | 404.2 (349.2)

8. Secondary Outcome: Dietary Cholesterol Intake
Description: Dietary cholesterol intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
milligrams
  Cholesterol (active) | 121.0 (82.3) | 143.2 (103.8)
  Cholesterol (control) | 113.1 (75.7) | 146.3 (112.9)

9. Secondary Outcome: Dietary Fiber Intake
Description: Dietary fiber intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
grams
  Fiber (active) | 3.2 (2.6) | 4.4 (3.9)
  Fiber (control) | 3.2 (2.6) | 4.9 (4.3)

10. Secondary Outcome: Dietary Iron Intake
Description: Dietary iron intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
milligrams
  Iron (active) | 2.9 (1.7) | 3.3 (2.5)
  Iron (control) | 2.5 (1.3) | 3.5 (2.4)

11. Secondary Outcome: Dietary Potassium Intake
Description: Dietary potassium intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
milligrams
  Potassium (active) | 606.4 (304.1) | 739.1 (470.5)
  Potassium (control) | 544.4 (222.9) | 808.6 (509.2)

12. Secondary Outcome: Dietary Sodium Intake
Description: Dietary sodium intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
milligrams
  Sodium (active) | 2045.5 (1215.1) | 2350.4 (1393.2)
  Sodium (control) | 1865.3 (1047.6) | 2255.8 (1376.1)

13. Secondary Outcome: Dietary Saturated Fat Intake
Description: Dietary saturated fat intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
grams
  Sat_Fat (active) | 14.5 (13.2) | 19.5 (11.5)
  Sat_Fat (control) | 13.6 (9.8) | 18.4 (12.3)

14. Secondary Outcome: Dietary Vitamin D Intake
Description: Dietary Vitamin D Intake was calculated across all food consumed during the ad lib buffet meal and summed to estimate total intake and compare between active and control conditions.
Time Frame: intake was assessed over a 30 minute meal
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
mcg
  Vit D (active) | 0.16 (0.22) | 0.25 (0.22)
  Vit D (control) | 0.16 (0.20) | 0.25 (0.30)

15. Secondary Outcome: Difference in Food Cravings
Description: Total score in the Food Cravings Questionnaire State (FCQ-State) after the vaping vs after the non-vaping condition. Fifteen items are rated on a 5-point Likert Scale (Strongly Disagree=1, Disagree=2, Neutral=3, Agree=4, Strongly Agree=5) with higher scores indicating higher food cravings. For a total score, all 15 items were summed together and higher scores indicate a higher intensity or craving to eat (Meule, 2020). The range for total scores is around 15-75.
Time Frame: The FCQ-State was administered about 30 minutes after either the vaping or non-vaping (control) condition and about ~20 minutes before the ad lib buffet meal.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vaping to Control Group | Control to Vaping Group
Number analyzed (Participants) | 18 | 16
units on a scale
  Total FCQ (active) | 49.8 (10.6) | 48.7 (8.4)
  Total FCQ (control) | 46.5 (12.3) | 52.2 (10.0)

ADVERSE EVENTS:
Time Frame: Data were collected following enrollment (screening/baseline visit) until completion of the final session or last date of contact with the participant (if withdrawn). The typical length of the study participation was approximately 2-4 weeks.
Description: At screening/baseline participants self-reported current physical symptoms and health conditions. Upon arrival to each study session, participants took a pre-session questionnaire to measure any changes in health since the previous in-person visit. Participants could also spontaneously report changes in health.
  Of note - the only AE observed for the Vaping to Control Group occurred during the Vaping (active) condition and was spontaneously reported.
Groups:
- Vaping to Control Group: Participants in this arm will undergo the vaping condition during the first visit and the control condition during the second visit.
  Please note, due to the way the arms/groups were described originally in clinicaltrials.gov, reporting for these outcomes is provided by condition order not by individual intervention or arm. Please see additional detail for the adverse event described above.
- Control to Vaping Group: Participants in this arm will undergo the control condition during the first visit and the vaping condition during the second visit.
  Please note, due to the way the arms/groups were described originally in clinicaltrials.gov, reporting for these outcomes is provided by condition order not by individual intervention or arm. Please see additional detail for the adverse event described above.
Arm/Group | Vaping to Control Group | Control to Vaping Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 1/18 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaping to Control Group (N=18) | Control to Vaping Group (N=16)
Dizziness (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT04219189/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT04219189/ICF_000.pdf